CLINICAL TRIAL: NCT05628844
Title: Uptake of Glucose and Phenylalanine From Continuous Enteral Nutrition in Healthy and Critically Ill Persons
Brief Title: Nutrient Uptake During Continuous Enteral Feeding
Status: Not yet recruiting | Type: Observational
Sponsor: Felix Liebau (Other Government)
Collaborators: Karolinska University Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Felix Liebau, Principal Investigator, Region Stockholm
Organization: Region Stockholm (Other Government)
Other Study IDs: 2022-04200-01
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Critical Illness
Keywords: Continuous enteral feeding; Gastric volume; Intestinal absorption; Enteral nutrition; Nutritional support
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: Healthy persons ≥ 18 yrs of age
  Interventions: Procedure: Continuous enteral feeding
- Critically ill patients: Critically ill patients ≥ 18 yrs of age admitted to the ICU
  Interventions: Procedure: Continuous enteral feeding

INTERVENTIONS:
Procedure: Continuous enteral feeding — Enteral nutrition by continuous infusion for 10 hrs at a dose corresponding to 25 kcal/kg body weight/day
  Other Names: Gastric ultrasound

SUMMARY:
Continuous enteral nutrition is used to feed patients in intensive care who are unable to eat normally. The goal of this observational study is to learn about the uptake of nutrients from feeding formula. The study method will first be applied in healthy persons to establish workability and normal values, then in patients in the intensive care unit to learn how nutrient uptake is affected by critical illness.

The main questions this study aims to answer are:

* what is the time course of uptake of phenylalanine (an amino acid) and glucose (a sugar) from enteral feeding formula given continuously over several hours
* what is the time course of the filling volume of the stomach during continuous enteral feeding

Participants receive feeding formula through a nasogastric feeding tube and blood samples are taken at short intervals to analyse uptake of nutrients into blood. Simultaneously, the filling volume of the stomach is measured by gastric ultrasound.

DETAILED DESCRIPTION:
Background

The investigators have previously studied the uptake of dietary isotope-labeled phenylalanine and plasma amino acid concentrations in critically ill patients and healthy subjects. During continuous feeding, uptake was unexpectedly found to be highly variable over time. Due to infrequent sampling, the time course of variability could not be modeled mathematically. Also, the underlying physiological mechanisms remain unclear, though it is hypothesized that gastric emptying is a major factor determining temporal variability.

The study here described is a follow-up that includes serial abdominal ultrasound studies to measure gastric emptying, additional indicators/tracers to determine more detail of uptake vs. digestion/transport/metabolism, and makes use of more frequent sampling to allow for detailed mathematical modeling of temporal variability.

Experimental protocol

ICU patients:

* Standard care and treatment as per clinical routines
* Pre-experiment ongoing nutrition for ≥ 6 hrs by nasogastric feeding tube or gastrostomy (not postpyloric)
* Bed rest during experiment as feasible

Healthy subjects

* Keep dietary and training habits for ≥ 2 days before experiment start
* Overnight fast
* Bed rest during experiment as feasible
* Nasogastric feeding tube
* Arterial line in radial or ulnar artery

Nutrition, sampling, measurements

* Experimental nutrition by continuous infusion for 10 hrs
* Infusion rate corresponding to 25 kcal/kg body weight/day (calculated including metabolizable tracers/indicators)
* Arterial blood sampling (à 1 ml) every 5 min in pilot study (may adjust to 10 or 15 min depending on results of pilot study)
* Serial abdominal ultrasound for determination of gastric volume (pilot study will determine how often)

Experimental nutrition

* Commercially available feeding formula for ICU use (Fresubin® HP Energy or similar) with added phenylalanine and glucose indicators
* Intrinsically labeled protein: 13C-L-phenylalanine intrinsically labeled milk protein
* Nonmetabolisable phenylalanine analogue: D-phenylalanine
* Free amino acid tracer: stable isotope-labeled phenylalanine tracer (2H5-L-Phe)
* Non-metabolizable glucose analogue: 3-O-Methyl-d-glucose (3-OMG)
* Free glucose tracer: isotope labeled D-glucose

Analyses

* arterial plasma amino acid and glucose tracers as above
* arterial plasma 3-OMG
* arterial plasma aminograms
* arterial plasma glucose, insulin, c peptide

ELIGIBILITY:
Inclusion Criteria (ICU patients):

- stable enteral nutrition of >80% of measured or calculated energy expenditure by nasogastric feeding tube or gastrostomy

Exclusion Criteria (ICU patients):

* enteral nutrition by postpyloric route such as jejunostomy or postpyloric tube
* remaining ICU stay expected < 12 hrs
* ongoing bleeding that requires surgery/intervention or transfusion of > 2 units red cells/24 hrs
* inability to use feeding tube or arterial line

Inclusion Criteria (healthy subjects):

- healthy volunteer

Exclusion Criteria (healthy subjects)

- any condition or medication affecting nutrition or metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ICU patients: patients admitted to an intensive care unit at Karolinska University Hospital
  Healthy subjects: volunteers from Stockholm metropolitan region
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Glucose and phenylalanine indicators | 0-10 hours
  Time series of isotopic and non-isotopic indicators of glucose and phenylalanine from enteral nutrition
Gastric volume | 0-10 hours
  Time series of gastric volume

SECONDARY OUTCOMES:
Plasma metabolites | 0-10 hours
  Time series of plasma aminograms, glucose, insulin and c peptide

CONTACTS AND LOCATIONS:
Overall Officials: Felix Liebau, MD PhD, Principal Investigator — Karolinska University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liebau F, Kiraly E, Olsson D, Wernerman J, Rooyackers O. Uptake of dietary amino acids into arterial blood during continuous enteral feeding in critically ill patients and healthy subjects. Clin Nutr. 2021 Mar;40(3):912-918. doi: 10.1016/j.clnu.2020.06.018. Epub 2020 Jun 30. PMID 32709553